CLINICAL TRIAL: NCT06659900
Title: Community Vital Signs (CVS): An Integrated Community-Based Approach to Identify Undiagnosed Hypertension in Nigeria
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Nigeria Nsukka (Other)
Responsible Party: Principal Investigator, Jennifer E DeVoe, MD DPhil, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IRB00027169
Record Dates: First submitted 2024-10-21; First posted 2024-10-26 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Hypertension
Keywords: Screening; Hypertension; Low-Middle Income; Nigeria; Implementation Science
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CORE (Arm A) (Experimental): CORE arm will use mHealth technologies to create data linkages with primary care facilities/providers, educational materials and a voucher for a medication starter kit
  Interventions: Other: CORE
- CORE PLUS (Arm B) (Experimental): CORE PLUS arm will use mHealth technologies to create data linkages with primary care facilities/providers, educational materials, a voucher for a medication starter kit PLUS support from a Community Health Advisor who will serve as a connector to primary care for HTN management and send reminder text messages.
  Interventions: Other: CORE Plus (+)

INTERVENTIONS:
Other: CORE Plus (+) — CORE PLUS intervention will use mHealth technologies to create data linkages with primary care facilities/providers, educational materials, a voucher for a medication starter kit PLUS support from a Community Health Advisor who will serve as a connector to primary care for HTN management and send reminder text messages.
  Arms: CORE PLUS (Arm B)
Other: CORE — CORE intervention will use mHealth technologies to create data linkages with primary care facilities/providers, educational materials and a voucher for a medication starter kit
  Arms: CORE (Arm A)

SUMMARY:
If detected early, hypertension (HTN) is treatable; yet, HTN screening rates are low and inequitable in Sub-Saharan Africa (SSA) leaving many people with undiagnosed HTN, especially in urban areas. Thus, it is a high priority to determine the acceptability, effectiveness, and sustainability of strategies to increase rates of BP screening and connections to care in SSA. The overarching goals of this project are to: 1. Adapt evidence-based implementation strategies - called community vital signs (CVS) strategies - to support BP screening and connections to care; 2. Implement the CVS strategies and assess acceptability, test their effectiveness in improving rates of BP screening and connections to care, and understand facilitators and barriers to their sustainability.

DETAILED DESCRIPTION:
Hypertension (HTN) is a leading modifiable risk factor for global cardiovascular disease and stroke morbidity and mortality. Nigeria, Africa's most populous country, has a high HTN burden. Evidence-based interventions (EBIs) for detection and initiation of treatment for HTN are not widely implemented in Nigeria. These EBIs include widely available BP screening (reaching all adults >18 years of age) to identify HTN early and connections to ongoing primary care for HTN management. In partnership with community and clinical stakeholders, we are currently adapting community-based strategies shown to be effective in increasing HIV screening and connections to care. The proposed adapted strategies - called community vital signs (CVS) strategies - will utilize community-based screenings, digital technologies, and supportive approaches to connect people to healthcare facilities, leveraging our practice-based research network of community clinics within the Model Innovation Research Centers created by the Nigeria Implementation Science Alliance. The study team will use the RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance) and EPIS (Exploratory, Preparation, Implementation, Sustainment) implementation science frameworks to guide the project.

Aim 1 / R61 Phase (Year 1): Engage stakeholders to refine and finalize the co-creation of CVS strategies aiming to increase rates of BP screening and connections to care in Nigeria. By the end of the R61 Phase, the study team will have final CVS strategies and will recruit, train, and conduct implementation readiness assessments at 12 community-based sites connected with 12 healthcare facilities in 12 Nigerian cities (2 in each of Nigeria's 6 regions).

R33 Phase (Years 2-5) Aim 2: Implement and assess CVS strategies aiming to increase rates of BP screening at all 12 study sites (n=24,000 participants). The study team will initiate quarterly, community-based BP screenings and evaluate using RE-AIM.

Aim 3: Implement and compare 2 different CVS strategies to make connections to primary care for those found to have high BP readings that meet HTN criteria at all study sites. The study team will conduct a nested, hybrid implementation-effectiveness type III trial using a parallel 2-arm cluster randomized design. Arm A (6 sites, n~3,000 participants): support connection to primary care by utilizing mHealth digital technologies with bidirectional sharing of BP data between community screening site and primary care clinic, coupled with a voucher for a medication starter kit (core strategies); Arm B (6 sites, n~3,000 participants): Core strategies plus community health navigators making handoffs to clinic and sending text messages (core+ strategies). This project promotes equitable access to HTN diagnosis and connections to care, especially in cities where HTN prevalence is highest.

It has the potential to significantly increase rates of early HTN detection and prevent the morbidity and mortality associated with the downstream effect of undiagnosed and uncontrolled HTN. It will provide evidence for scale-up of interventions to support self-management of non-communicable chronic diseases in Nigeria and other low- and middle-income countries.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>= 18 years of age)

Exclusion Criteria:

* Children (< 18 years of age)
* prisoners
* neonates
* adults lacking capacity
* taking antihypertensive medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24000 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Reach of intervention | Any point during the 24 month intervention period
  the rate of participants who were offered BP screening by those who received BP screening
Effectiveness of Intervention | Any point during the 24 month intervention period
  Proportion of patients who were screened for HTN and met HTN threshold who were connected to care. This will be a site-level analysis using GEE models.
Adoption of intervention by intervention sites | Any point during the 24 month intervention period
  Adoption will be measured using community-observations and period reflections from the site research coordinators who conduct the intervention. The investigators will assess how well-informed community members feel about the purpose of BP screenings, the need to connect to care for ongoing HTN management, the use of tools provided by the team, and if they deviated from the study protocol to achieve the goals of the intervention.
Fidelity to the Implementation of the Intervention | Years 2-4
  Longitudinal data from the Implementation Climate Measure, a survey used to assess implementation readiness, will be summarized within an across intervention sites and GEE models will be used to evaluate changes across time.
Maintenance of Intervention | Years 2-5
  Proportion of patients who were screened at baseline who return for a repeat screening. This will be assessed within and across all study sites.

SECONDARY OUTCOMES:
Impact of intervention on diagnoses of HTN | Years 2-5
  Percent of people referred for care who get diagnosed with HTN and begin treatment on appropriate medications
Cost Effectiveness | Years 1-5
  Mean total annual costs for years 1-5, including intervention preparation and implementation by site and overall.
Impact of intervention on BP | 12 and 24 months after enrollment
  Percent of people referred for care who have improved BP over time, measured at quarterly screening

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nigeria, Nsukka, Enugu, Nigeria